CLINICAL TRIAL: NCT02590770
Title: Gaze Contingent Feedback in Treatment of SAD
Brief Title: Gaze Contingent Feedback in Social Anxiety Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Yair Bar-Haim, Professor of Psychology and Neuroscience School of Psychological Sciences Sagol School of Neuroscience Tel Aviv University, Tel Aviv University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAUSAD
Record Dates: First submitted 2015-10-27; First posted 2015-10-29 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: Phobia, Social
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- gaze-contingent (Active Comparator): attention modification: participants will receive gaze-contingent feedback according to their viewing patterns
  Interventions: Behavioral: attention modification
- non-gaze contingent (Placebo Comparator): Placebo: participants will receive non-gaze-contingent feedback according to their viewing patterns
  Interventions: Other: Placebo

INTERVENTIONS:
Behavioral: attention modification — participants will receive gaze-continent feedback according to their viewing patterns
  Arms: gaze-contingent
Other: Placebo — participants will receive non-gaze-continent feedback unrelated to their viewing patterns
  Arms: non-gaze contingent

SUMMARY:
The purpose of this study is to determine whether giving gaze-contingent feedback is an effective attention modification procedure, helping in the treatment of social anxiety disorder (SAD)

DETAILED DESCRIPTION:
The study examines giving social anxious participants gaze-contingent feedback as a novel attention training procedure. Half of the participants will receive contingent feedback while the other half would receive non-contingent "placebo" feedback.

ELIGIBILITY:
Inclusion Criteria:

* A signed consent form
* Men and women between the ages of 18 and 60.
* Meeting a current diagnosis of Social Anxiety Disorder (SP) according to the DSM-IV
* A minimum of a 1-year duration of SP
* SP as the primary diagnosis: In cases of co-morbidity, SP will be deemed as the most distressing and clinically significant condition among the co-morbid disorders
* Stable pharmaco-therapy: Participants receiving a pharmacological treatment who are taking a stable medication for at least 3 months before the beginning of the procedure.

Exclusion Criteria:

* Psychotic episode in the past or the present time.
* Co-morbidity with any neurological disorder (i.e., epilepsy, brain injury).
* Another psychotherapeutic treatment during the study.
* Usage of neuroleptic medication.
* Change in medication status during the study.
* Substantial usage of drugs or alcohol in the present time.
* Poor judgment capacity (i.e., children under 18 and special populations).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-10; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline - the Liebowitz Social Anxiety Scale - Diagnostic Interview scores | post treatment (1 week after treatment completion) and 3-month follow up
  The LSAS is a 24-item scale, each item corresponding to a situation selected on the basis of clinical experience. Each item is rated on a severity scale ranging from 0 to 3 with regard to the passing week, measuring separately two components of social anxiety, specifically, fear/anxiety and avoidance of social interaction and performance situations. Although the assessor may request and ask for further detail and adjust the rating based on clinical experience, this option is not often exercised, and inter-rater agreement is not considered to be a relevant concern. It has been shown to have strong psychometric properties, including high internal consistency, strong convergent and discriminative validity and high test-retest reliability.

SECONDARY OUTCOMES:
Change from baseline - the Social Phobia Inventory scores | post treatment (1 week after treatment completion) and 3-month follow up
  This is a 17-item self-report measure of social anxiety evaluating fear, avoidance and physiological discomfort. Each item is rated on scale ranging from 0 to 4 with a possible total score of 68. The SPIN has been used in clinical and nonclinical samples and its psychometric properties have been found to be sound.

OTHER OUTCOMES:
changes in the Mini-International Neuropsychiatric Interview (M.I.N.I) diagnosis | post treatment (1 week after treatment completion)
  a structured diagnostic interview for DSM - IV and ICD-10 psychiatric disorders, which takes approximately 20 min to administer and is a valid and time-efficient alternative to the SCID-P and CIDI.

CONTACTS AND LOCATIONS:
Overall Officials: Yair Bar-Haim, PhD, Principal Investigator — Tel Aviv University
Locations (1):
- Tel-Aviv University, Tel Aviv, Israel

REFERENCES:
- [Derived] Lazarov A, Pine DS, Bar-Haim Y. Gaze-Contingent Music Reward Therapy for Social Anxiety Disorder: A Randomized Controlled Trial. Am J Psychiatry. 2017 Jul 1;174(7):649-656. doi: 10.1176/appi.ajp.2016.16080894. Epub 2017 Jan 20. PMID 28103714